CLINICAL TRIAL: NCT04013165
Title: Effectiveness of a Village-based Intervention for Depression in Community-dwelling Older Adults: a Randomized Controlled Pilot Study
Brief Title: Village-based Intervention for Late-life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VILLD
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-05

CONDITIONS: Depression
Keywords: Old-aged; Community-based intervention; Late-life depression; Suicide
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Intervention Model Description: A community-based randomized controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active control (Active Comparator): Usual care of the Community Mental Health Service
  Interventions: Behavioral: Active control
- Village-based intervention (Experimental): Individual-based case management + group-based program
  Interventions: Behavioral: Village-based intervention

INTERVENTIONS:
Behavioral: Active control — Control group received usual care of the Community Mental Health Service, consisted of case management for high-risk older adults and referral to psychiatric services.
  Arms: Active control
Behavioral: Village-based intervention — 1. Individual-based case management was conducted both by healthy community dwellers (local committee) and Community Mental Health Service (CMHS) team based on risk-stratification for depression in older adults. Local committee-guided care was performed after matching a healthy dweller with 4-5 older neighbors included in risk groups. They visited the matched older individuals as often as possible at least once a week using a mood sticker. The CMHS team also conducted a separate case management for older adults with risk-stratified protocols; the higher the risk of suicide, the more intensive was the management, which could include frequent face-to-face visits. High-risk individuals were also referred to the psychiatric service, if deemed necessary.
  2. Group-based program was comprised of weekly eight sessions, which were mainly consisted of programs enhancing interpersonal network and group cohesion, and were open to all community-dwelling older adults.
  Arms: Village-based intervention

SUMMARY:
Investigators aimed to examine the feasibility and effectiveness of a village-based multilevel intervention for late-life depression. Two small rural villages in rural South Korea were selected as the intervention group and active control. All older adults living in the two villages were included in the intervention program or received standard CMHS care, and the effectiveness of the program was examined using representative samples from both groups.

DETAILED DESCRIPTION:
OBJECTIVES: To examine the feasibility and effectiveness of a village-based multilevel intervention for late-life depression, focusing on strengthening the autonomy of village-dwellers with help from the community mental health service (CMHS).

DESIGN: A community-based randomized trial with participants (all village-dwellers) assigned to two parallel programs: intervention program or the CMHS's usual care.

SETTING: Two small villages in a rural area of South Korea

PARTICIPANTS: All older adults (aged ≥65 years) living in the two villages were included in the intervention or the CMHS's usual care, and the effectiveness of the program was examined using representative samples who were age- and sex-stratified randomly selected from both groups.

INTERVENTION: A 12-week intervention was comprised of individual-based risk-stratified case management and group-based activities.

MEASUREMENTS: The Korean version of Geriatric Depression Scale-Short form (SGDS-K) was used as the primary outcome while depressive episodes, suicidal ideation/plans/attempts, social network, functional status, and global cognitive function were measured as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All community-dwelling older adults, aged 65 years and over

Exclusion Criteria:

* Subjects who had significant sensory deficits or medical illnesses that would substantially restrict the delivery of the assessment were excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Korean version of the short form of Geriatric Depression Scale (SGDS-K) after intervention | baseline, after intervention (up to 24 weeks)
  The SGDS-K was developed for evaluating depressive symptoms of older adults; higher score means to have more depressive symptoms (lowest 0 - highest 15)

SECONDARY OUTCOMES:
Incidental depressive episode after intervention | baseline, after intervention (up to 24 weeks)
  Major or minor depressive episode was diagnosed based on the Diagnostic and Statistical Manual of Mental Disorders, the fourth edition (DSM-IV) using a structured clinical interview, the Korean Version of the Composite International Diagnostic Interview (K-CIDI)
Incidental suicidal ideation, plans, or attempts after intervention | baseline, after intervention (up to 24 weeks)
  Multisite Intervention Study on Suicidal Behaviours (SUPRE-MISS) was used to assess of having suicidal ideation, plans, or attempts.
Changes from baseline Korean version of Lubben Social Network Scale (K-LSNS) after intervention | baseline, after intervention (up to 24 weeks)
  The Lubben Social Network Scale (LSNS) was developed for evaluating older adults' social interaction with their relatives and friends; higher score means to have stronger social network (lowest 0 - highest 50).
Changes from baseline Seoul-Instrumental Activities of Daily Living (S-IADL) after intervention | baseline, after intervention (up to 24 weeks)
  Seoul-Instrumental Activities of Daily Living (S-IADL) was developed to assess elderly person's instrumental everyday activities; higher score means to have worse daily function (lowest 0 - highest 45).
Changes from baseline Korean version of the Mini-Mental State Examination (MMSE-KC) after intervention | baseline, after intervention (up to 24 weeks)
  Mini-Mental State Examination in the Korean version of the CERAD assessment packet (MMSE-KC) is a well-known screening tool for global cognitive function that measures orientation, language (repetition, naming, reading and writing), concentration, constructional praxis, and memory; higher score means to have better global cognitive function (lowest 0 - highest 30).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh IM, Cho MJ, Hahm BJ, Kim BS, Sohn JH, Suk HW, Jung BY, Kim HJ, Kim HA, Choi KB, You DH, Lim AR, Park IO, Ahn JH, Lee H, Kim YH, Kim MR, Park JE. Effectiveness of a village-based intervention for depression in community-dwelling older adults: a randomised feasibility study. BMC Geriatr. 2020 Mar 4;20(1):89. doi: 10.1186/s12877-020-1495-2. PMID 32131745